CLINICAL TRIAL: NCT01376505
Title: Phase I Active Immunotherapy Trial With a Combination of Two Chimeric (Trastuzumab-like and Pertuzumab-like)Human Epidermal Growth Factor Receptor 2 (HER-2) B Cell Peptide Vaccine Emulsified in ISA 720 and Nor-MDP Adjuvant in Patients With Advanced Solid Tumors
Brief Title: Vaccine Therapy in Treating Patients With Metastatic Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Robert Wesolowski (Other)
Responsible Party: Sponsor-Investigator, Robert Wesolowski, Principal Investigator, Ohio State University Comprehensive Cancer Center
Organization: Ohio State University Comprehensive Cancer Center (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OSU-09138; NCI-2011-00920 (Registry Identifier: Clinical Trial Reporting Program)
Record Dates: First submitted 2011-06-09; First posted 2011-06-20 (Estimated); Last update posted 2023-09-15 (Actual); Status verified 2023-09

CONDITIONS: Malignant Solid Tumour; Breast Cancer; Malignant Tumor of Colon; GIST; Ovarian Cancer
Keywords: Vaccine Therapy
MeSH Terms: conditions — Breast Neoplasms; Colonic Neoplasms; Ovarian Neoplasms | interventions — CHP-HER2 vaccine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- HER-2 Vaccine (Experimental): combination of MVF-HER-2 (597-626) and MVF-HER-2 (266-296) emulsified with nor-MDP and ISA 720
  This escalation arm has completed. The trial has moved on to the extension arm
  Interventions: Biological: HER-2 vaccine
- EXTENSION HER-2 Vaccine at OBD (Experimental): Combination of MVF-HER-2 (597-626) and MVF-HER-2 (266-296) emulsified with nor-MDP and ISA 720 at dose level cohort 2
  This extension arm is ongoing
  Interventions: Biological: Extension HER-2 vaccine trial at OBD

INTERVENTIONS:
Biological: HER-2 vaccine — Three intramuscular (IM) injections (separated by 21 days) of a mixture of two peptides {MVF-HER-2(597-626) and MVF-HER-2 (266-296)} vaccine emulsified with nor-MDP in ISA 720 vehicle. Increasing doses of the combined vaccine preparation emulsified with nor-MDP (0.025) mg and Montanide ISA 720 will be administered in a final volume of 1.0 ml. Starting at dose level 1, 1.0mg of each peptide will be used for vaccination. In increasing dosing cohorts 1.5mg, 2.0mg and 2.5mg will be used. Patients may also receive 6 months booster shots.
  Other Names: Synthetic peptides of HER-2 comprising B cell epitopes with a Promiscuous T cell epitope of Measles Virus.
  Arms: HER-2 Vaccine
Biological: Extension HER-2 vaccine trial at OBD — Three intramuscular (IM) injections (separated by 21 days) of a mixture of two peptides {MVF-HER-2(597-626) and MVF-HER-2 (266-296)} vaccine emulsified with nor-MDP in ISA 720 vehicle. The dose level has been determined to be cohort 2. The combined vaccine preparation consists of 1.5mg of each of the HER-2 vaccine emulsified with nor-MDP (0.025) mg and Montanide ISA 720 will be administered in a final volume of 1.0 ml. Patients may also receive 6 months booster shots.
  Arms: EXTENSION HER-2 Vaccine at OBD

SUMMARY:
This phase I trial studies the side effects and best dose of vaccine therapy in treating patients with metastatic solid tumors. Vaccines made from antibodies and peptides combined with tumor cells may help the body build an effective immune response to kill tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To perform early phase clinical trial assessing safety and clinical toxicity of immunization, and as well as to establish an optimal biological dose (OBD) of combination vaccines with n-muramyldipeptide derivative (nor-MDP) as adjuvant emulsified in Montanide (ISA 720).

II. To establish whether an OBD of two combination vaccines is achieved. III. To measure both humoral and cellular immune responses including the specificity, class and kinetics of anti-human epidermal growth factor receptor-2 (HER-2) peptide.

IV. To evaluate whether the combination of HER-2 epitopes show therapeutic benefit, provide synergistic and/or additive effects and to enumerate mechanisms of action.

SECONDARY OBJECTIVES:

I. To collect and analyze post-immune sera and peripheral blood cells for additional six months post the last injection.

II. To document any clinical responses that may occur.

OUTLINE: This is a dose-escalation study.

Patients receive a HER2/neu peptide vaccine comprising measles virus epitope MVF-HER-2 (266-296) and MVF-HER-2 (597-626) emulsified with nor-MDP in ISA 720 intramuscularly (IM) on day 1. Treatment repeats every 21 days for up to 3 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days.

OUTLINE: EXTENSION TRIAL AT OBD

The dose-escalation (4 cohorts) has successfully completed with the accrual of 24 patients and the Optimum biological dose (OBD) has been determined as the dose at cohort level 2.

The next phase of the study progresses directly into an extension trial at the OBD. 12 patients will be accrued at that level. The extension cohort will be open to only HER-2 and/or EGFR overexpressing cancers. Patients (all gastrointestinal,ovarian and breast must have received no more than three prior cytotoxic chemotherapy regimens in the last two years after standard therapy. Patients (breast, ovarian and gastrointestinal cancers) must have received no more than three prior cytotoxic chemotherapy regimens in the last two years after standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Must have histologically confirmed metastatic solid tumor; the malignancy should be considered incurable using standard treatment
* Patients are not required to have HER-2 over-expression to be on this study
* If the patient has had HER-2 expression measured prior to enrollment, the report alone will be accepted
* If the patient has not had HER-2 expression measured prior to enrollment on this study tumor tissue blocks and/or freshly isolated tissue must be available for determination of HER-2 expression
* Patients are not required to have epidermal growth factor receptor (EGFR) over-expression to be on this study
* If the patient has had EGFR expression measured prior to enrollment, the report alone will be accepted
* If the patient has not had EGFR expression measured prior to enrollment on this study tumor tissue blocks and/or freshly isolated tissue must be available for determination of EGFR expression
* Patients with prior history of treated brain metastases who are off steroids and have stable metastatic brain disease for at least 3 months are eligible
* Patients must be ambulatory with an Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2

  * White blood cells > 3500/mm^3
  * Platelet count > 100,000/mm^3
  * Serum bilirubin < 1.5 mg %, regardless of whether patients have liver involvement secondary to tumor
  * Alanine aminotransferase (ALT) must be < 2 times upper limit of normal
  * Creatinine < 1.5 mg/dL or calculated creatinine clearance > 60 mL/min
* Patients will be tested for reactivity to a panel of four common microbial skin test antigens: candida, trichophyton, intermediate strength purified protein derivative (PPD), and tetanus toxoid; determination of patient eligibility for this trial will proceed independently of these skin test results; patients who have previously been tested for these antigens but were excluded from participation in the trial due to non-reactivity may be considered as eligible provided that all other eligibility criteria are met
* Patients must be at least 4 weeks past any prior surgery, cytotoxic, chemotherapy, other immunotherapy, hormonal therapy, or radiation therapy; patients having been treated with monoclonal antibodies may enter the trial after a specified period of time (2 times the mean half life of the agent); patients must have recovered from any toxicity of prior therapy prior to enrolling on study except for neuropathy where patients need to recover to less than grade 2
* Women of child-bearing potential must not be pregnant and must have a negative pregnancy test; men and women must agree to practice effective contraception while on this study
* Patients must obtain a base line Echocardiogram or multi gated acquisition scan (MUGA) and require the left ventricular ejection fraction to be within normal limits (or 50% or higher)
* Ability to understand and the willingness to sign a written informed consent document; the patient must be aware that his/her disease is neoplastic in nature and willingly consent after being informed of the procedure to be followed, the experimental nature of the therapy, alternatives, potential benefits, side-effects, risks, and discomforts

Exclusion Criteria:

* Patients with ICH of 0
* Patients on targeted therapies, such as Cycline Dependent Kinase (CDK) 4/6 or mammalian target of rapamycin (mTOR) inhibitors in combination with endocrine therapy.
* Patients who are {MVF-HER-2(266-296) and MVF-HER-2 (597-626)} immediate hypersensitivity skin test positive
* Patients who have evidence of active infection that requires antibiotic therapy; patients must have been off antibiotic treatment for at least 3 weeks prior to initiating treatment and must be confirmed to be clear of the infection; if patient develops an infection requiring antibiotic treatment while on the treatment portion of the study patients will be treated for the active infection with antibiotics and will resume vaccine treatment when the infection is healed
* Patients with known active human immunodeficiency virus (HIV), hepatitis A, hepatitis B, or hepatitis C infection
* Patients with serious cardiopulmonary disorders, including congestive heart failure, symptomatic coronary artery disease, serious cardiac arrhythmia, and symptomatic chronic obstructive pulmonary disease or patients with other serious uncontrolled medical diseases
* Patients who require or likely to require corticosteroids or other immunosuppressives for intercurrent disease are NOT eligible
* Splenectomized patients
* Autoimmune diseases including rheumatoid arthritis, systemic lupus erythematosus, scleroderma, polymyositis dermatomyositis, or a vasculitic syndrome
* Patients who have developed anaphylactic responses to other vaccines
* History of congestive heart failure, coronary artery disease and myocardial infarction; active or unstable cardiovascular disease or cardiac disease requiring drug or device intervention

ADDITIONAL KEY ELIGIBILITY CRITERIA FOR EXTENSION & EXPANSION COHORT:

* Histologically documented metastatic or unresectable breast, ovarian and gastrointestinal cancers
* Progressive disease after at least one line of standard therapy
* Patients must have received or refused first line standard systemic therapy for their metastases (if applicable)
* Patients (pancreatic and esophageal cancers) must have received no more than two prior cytotoxic chemotherapy regimens in the last two years after standard therapy. Patients (breast and gastrointestinal cancers) must have received no more than three prior cytotoxic chemotherapy regimens in the last two years after standard therapy.
* Measurable disease, defined as ≥ 1 lesions that can be accurately measured in ≥ 1 dimensions as ≥ 20 mm with conventional techniques or as ≥ 10 mm with spiral CT scan
* Disease that is amenable to biopsy and be willing to undergo tumor biopsy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Actual)
Dates: Start 2011-06-21 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

PRIMARY OUTCOMES:
Type and duration of immune response measured over time to repeat vaccine administration | up to 6 months
  Immune response will be defined by Enzyme-linked immunosorbent assay (ELISA), Flow cytometry, T-cell proliferation and cytokine. The magnitude of antibody levels will be assessed to the vaccine and HER-2 over-expressing cells (e.g.,BT474). Lymphoproliferative responses will be assessed by a non radioactive cell proliferation assay Bioplex human isotyping kit will be used to assess antibody types and cytokine profiles.
Clinical benefit will be assessed | up to 6 months
  Will re-evaluate disease status with tumor markers and RESIST criteria,or full evaluation upon development of new symptoms

SECONDARY OUTCOMES:
Evaluation of safety and toxicity at regular intervals by NCI common toxicity criteria (CTCAE v 4.0) | up to 6 months
  Safety will be defined if patients are able to receive all 3 vaccinations without dose-limiting toxicity (DLT), any incidence of grade 3 hematologic and non-hematologic toxicity or any incidence of Grade 4 toxicity. The development of a positive skin test to the vaccine immediate hypersensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Robert Wesolowski, MD, Principal Investigator — Ohio State University
Locations (1):
- Ohio State University Medical Center, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bekaii-Saab T, Wesolowski R, Ahn DH, Wu C, Mortazavi A, Lustberg M, Ramaswamy B, Fowler J, Wei L, Overholser J, Kaumaya PTP. Phase I Immunotherapy Trial with Two Chimeric HER-2 B-Cell Peptide Vaccines Emulsified in Montanide ISA 720VG and Nor-MDP Adjuvant in Patients with Advanced Solid Tumors. Clin Cancer Res. 2019 Jun 15;25(12):3495-3507. doi: 10.1158/1078-0432.CCR-18-3997. Epub 2019 Feb 25. PMID 30804020
- See also: Jamesline — http://cancer.osu.edu